CLINICAL TRIAL: NCT06159140
Title: Small Vessel Diseases: Ultra-realistic Microstructure Computational Model to Refine Individual Treatment
Acronym: SUMMIT-WP3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DR220256-SUMMIT; DR220256 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-11-24; First posted 2023-12-06 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Small Vessel Disease
Keywords: MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental): MRI and neuropsychological evaluation
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — In vivo MRI

SUMMARY:
Small vessel disease (SVD) accounts for 25% of strokes and is the second most common cause of dementia after Alzheimer's disease. Unlike other causes of stroke, SVD manifests itself years before the stroke by the accumulation of tissue damage. Although heterogeneous, these lesions appear on Magnetic Resonance Imaging (MRI) as white matter hypersignals (WMH). In this context, the ANR SUMMIT project will characterize these lesions in vivo to develop new markers in the early stages of stroke. It is subdivided into 4 work packages, the third one being promoted by CHRU de Tours.

ELIGIBILITY:
Inclusion Criteria:

Prior Enrollement in Tours body donation program Age ≥ 82 years Able to remain supine in the MR scanner for acquisition (duration 60-minutes) Affiliation to social security Informed and written consent

Exclusion Criteria:

Contraindications to body donation, especially infectious disease (VIH, HBV…) Contraindications to MRI

Ages: 82 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
In vivo and ex vivo MRI measures data | baseline
  We will compare In vivo data: 20 MR datasets, 20 quantitative SUMMIT maps (predicted microstructure)
  Ex vivo data :
  * 3 very high-resolution MR datasets and derived quantitative microstructural maps
  * 18 brain samples: scanned at 17.2T by the Neurospin partner and processed with the SUMMIT method to obtain high-resolution quantitative microstructural maps
  * these 18 samples will be processed to get ground truth histological 3D volumes (Mircen partner).
  Maps of the microstructure parameters obtained from MRI (in and ex vivo) and the SUMMIT method will be quantitatively compared to histological data.
  This will validate the SUMMIT method at clinical (in vivo) and mesoscopic resolution (ex vivo).

SECONDARY OUTCOMES:
FLAIR and SUMMIT maps (MRI evaluation) | baseline
  In vivo FLAIR and SUMMIT maps.
Scores at neuropsychological evaluation | baseline
  Scores at neuropsychological evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- UHT of Tours, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided